CLINICAL TRIAL: NCT03822754
Title: A Randomized, Double-blind, Controlled Clinical Trial to Evaluate the Immunogenicity and Safety of Sabin Inactivated Poliovirus Vaccine (Vero Cell) in a '1+2' Sequential Schedule With Bivalent Oral Poliovirus Vaccine in 2-month-old Infants
Brief Title: A Clinical Trial to Evaluate the Immunogenicity and Safety of sIPV in a '1+2' Sequential Schedule With bOPV in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-sIPV-3001-1
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Poliomyelitis
Keywords: Sabin strain; Inactivated poliovirus vaccine; poliomyelitis; safety; immunogenicity; infant; sequential schedule
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): sIPV-bOPV-bOPV vaccination schedule
  Interventions: Biological: sIPV-bOPV-bOPV vaccination schedule
- Control Group (Active Comparator): wIPV-bOPV-bOPV vaccination schedule
  Interventions: Biological: wIPV-bOPV-bOPV vaccination schedule

INTERVENTIONS:
Biological: sIPV-bOPV-bOPV vaccination schedule — Single intramuscular injection of the experimental sIPV (0.5 ml) on Day 0, following two doses of bOPV (0.1 ml) on Day 30 and Day 60 respectively. The investigational Sabin strain inactivated poliovirus vaccine (Vero cell)(sIPV) was manufactured by Sinovac Vaccine Technology Co., Ltd. The poliovirus (Live) vaccine type I & type III (Human Dipoid cell) ( bOPV) was manufactured by Beijing Bio-institute Biological Products Co., Ltd.
  Arms: Experimental Group
Biological: wIPV-bOPV-bOPV vaccination schedule — Single intramuscular injection of the control wIPV (0.5 ml) on Day 0, following two doses of bOPV (0.1 ml) on Day 30 and Day 60 respectively.The control wild strain inactivated poliovirus vaccine (wIPV) was manufactured by SANOFI PASTEUR S.A. The poliovirus (Live) vaccine type I & type III (Human Dipoid cell) ( bOPV) was manufactured by Beijing Bio-institute Biological Products Co., Ltd.
  Arms: Control Group

SUMMARY:
The purpose of this phrase III clinical trial is to evaluate the immunogenicity and safety of Sabin Inactivated Poliovirus Vaccine (Vero cell) in a '1+2' sequential schedule with bivalent oral poliovirus vaccine in 2-month-old infants

DETAILED DESCRIPTION:
This study is a randomized, double-blind, active-controlled phrase III clinical trial. The purpose of this study is to evaluate the immunogenicity and safety of sIPV manufactured by Sinovac Vaccine Technology Co., Ltd in a '1+2' sequential schedule with bOPV in 2-month-old infants. 240 infants aged between 60-90 days will be randomly assigned into experimental group or control group in the ratio 1:1. The experimental group received sIPV-bOPV-bOPV vaccination schedule at one month doses interval (i.e., month 0, 1, 2), and the control group received wIPV-bOPV-bOPV vaccination schedule at one month doses interval (i.e., month 0, 1, 2). The control wIPV was manufactured by SANOFI PASTEUR S.A.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 60-90 days old;
* Healthy volunteers who fulfill all the required conditions for receiving the investigational vaccine as established by medical history and clinical examination and determined by investigators;
* Proven legal identity;
* Participants or guardians of the participants should be capable of understanding the written consent form, and such form should be signed prior to enrolment;
* Complying with the requirement of the study protocol;

Exclusion Criteria:

* Prior vaccination with Poliovirus Vaccine;
* History of allergy to any vaccine, or any ingredient, excipients and Gentamycin Sulfate of the vaccine, or serious adverse reaction(s) to vaccination, such as urticaria, dyspnea, angioneurotic edema, abdominal pain, etc;
* Congenital malformation, developmental disorders, genetic defects, or severe malnutrition;
* Autoimmune disease or immunodeficiency/immunosuppressive;
* Severe/uncontrollable nervous system disease (epilepsy, seizures or convulsions) or mental illness;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) prior to study entry;
* Blood product prior to study entry;
* Any other investigational medicine(s) within 30 days prior to study entry;
* Any live attenuated vaccine within 14 days prior to study entry;
* Any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Axillary temperature > 37.0 °C;
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators;

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
The difference between experimental group and control group of type I,III neutralizing antibody seroconversion rate after primary immunization. And the lower limit of 95% confidence intervals of the difference value. | 30 days
  Subjects whose pre-immune antibody level < 1:8 and post-immune antibody level ≥ 1:8, or those whose pre-immune antibody level ≥ 1:8 and the increase of post-immune antibody level ≥ 4 folds are considered seroconverted. Primary vaccination schedule: 3 doses with one month interval between doses (i.e., month 0, 1, 2).

SECONDARY OUTCOMES:
The incidences of solicited adverse events (AEs) within 7 or 14 days after each dose of each group. | 7 days or 14 days
  Solicited AEs occurred within 7 days (for sIPV/wIPV) or 14 days（for bOPV） after each injection will be collected.
The incidence of unsolicited AE within 30 days after each dose of each group. | 30 days
  Unsolicited AEs occurred within 30 days after each injection will be collected.
Incidence of serious adverse events (SAEs) during the period of safety monitoring. | 30 days.
  SAEs during the period of safety monitoring will be collected.
Type I,II and III neutralizing antibody positive rate of each group after primary immunization | 30 days
  Subjects whose post-immune antibody level ≥ 1:8 are considered antibody positive. Primary vaccination schedule: 3 doses with one month interval between doses (i.e., month 0, 1, 2).
Type I,II and III post-immune geometric mean titer (GMT) of each group after primary immunization. | 30 days
  GMT of each group after primary immunization
Type I,II and III post-immune geometric mean fold increase (GMI) of each group after primary immunization. | 30 days
  The GMI is the increase of post-immune GMT from pre-immune GMT.

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Guanyun Center for Disease Control and Prevention, Lianyungang, Jiangsu, China